CLINICAL TRIAL: NCT01374789
Title: PURO - An Open-label, Randomised, Multicentre, Phase II Study to Evaluate the Efficacy of Chemotherapy With Gemcitabine and Cisplatin in Combination With the EGF Receptor Antibody Panitumumab (GemCisP) Versus GemCis in the First-line Therapy of Locally Advanced/Metastatic Urothelial Carcinoma in Patients With Wild-type HRAS
Brief Title: PURO Panitumumab in Combination With Gemcitabine/Cisplatin in Advanced Urothelial Cancer
Acronym: PURO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to insufficient recruitment.
Sponsor: WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Collaborators: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WiSP_AG48; 2009-015119-42 (EudraCT Number); GMIHO-007/2008 (Other: GMIHO mbh)
Record Dates: First submitted 2011-03-30; First posted 2011-06-16 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (GemCis + Panitumumab) (Experimental): gemcitabine + cisplatin + panitumumab
  Interventions: Drug: GemCis + Panitumumab
- Arm B (GemCis) (Active Comparator): gemcitabine + cisplatin
  Interventions: Drug: GemCis

INTERVENTIONS:
Drug: GemCis + Panitumumab — Gemcitabine: 1250 mg/m², day 1 and 8, i.v., q3 Cisplatin: 70 mg/m², day 2, i.v., q3 Panitumumab 9 mg/kg/body weight, i.v., day 1,q3
  Other Names: Vectibix (Panitumumab)
  Arms: Arm A (GemCis + Panitumumab)
Drug: GemCis — Gemcitabine: 1250 mg/m², day 1 and 8, i.v., q3 Cisplatin: 70 mg/m², day 2, i.v., q3
  Arms: Arm B (GemCis)

SUMMARY:
The primary objective of the study is to assess the efficacy of the combination consisting of gemcitabine/cisplatin and panitumumab in patients with urothelial carcinoma and wild-type HRAS (non-mutated status). The progression-free survival rate at 12 months will be compared to expectations derived from historical data, which are verified by a randomised control group without the antibody.

DETAILED DESCRIPTION:
Mutation of ras oncogenes is frequently observed in human tumours and occurs in approximately 30% of all cancer types. Frequent mutation "hot spots" occur in codon 12 (glycine to valine), codon 13 (glycine to cysteine) and codon 61 (glutamine to arginine, lysine and leucine) (Bonner et al. 1993, Levesque et al. 1993). Point mutations in ras genes result in blockade of intrinsic GTPase activity, the physiological mechanism that switches off ras GTPases. The consequence is persistent up-regulation of the signal pathway and increased cell proliferation. The first HRAS mutation in association with bladder cancer was described during establishment of the human urinary bladder carcinoma cell line T24. In further studies, a research group led by Fitzgerald was able to demonstrate that HRAS gene mutations were present in the urine sediment of up to 44% of patients with urinary bladder cancer (Fitzgerald et al. 1995).

Viola et al. subsequently investigated whether an increased mutation rate is accompanied by increased expression of ras proteins in bladder cancer. It was shown that there is indeed increased expression of ras proteins in dedifferentiated tumours and carcinomas in situ, whereas highly differentiated tumours do not exhibit this rate of expression (Viola et al. 1985).

At present, there is no clinical evidence, that the findings of an obvious lack of activity of EGFR antibodies in colorectal cancer with RAS-related mutations, is likewise valid in urothelial carcinoma. However, as it is the aim of this study to detect a first signal of activity in this type of cancer, and the chance of missing such evidence in a phase II trial with limited patient numbers is high anyway, it seems sensible, not to miss this opportunity of "enrichment". In case of a clearly positive signal of efficacy in the present trial, a subsequent phase II study may focus on HRAS mutated tumors.

Overexpression of the EGF receptor in bladder cancer has been described by many research groups (Colquhuon & Mellon, 2002) and is associated with an advanced stage of the tumour, progression of the tumour and a poor clinical prognosis. The EGFR antibody cetuximab (Erbitux®) has been investigated in a human urothelial carcinoma cell line and in a mouse model with human bladder carcinoma. Cetuximab was found to inhibit tumorigenesis and metastatic progression in vivo and in vitro by means of suppression of angiogenesis and simultaneous induction of apoptosis (Perotte et al., 1999; Inoue et al., 2000). Similar results have also been reported in urothelial carcinoma for the tyrosine kinase inhibitor gefitinib (Villares et al., 2007, Shrader et al., 2007).

There are currently two on-going studies of cetuximab in metastatic bladder cancer: a randomised phase II study of first-line treatment with Gemcitabine and Cisplatin +/- Erbitux (NCT00645593) and a randomised phase II study of second-line treatment with Erbitux +/- Paclitaxel (NCT00350025).

The HRAS mutation rate in urothelial carcinoma is approximately 40%. The primary objective of the study is to assess the efficacy of the combination consisting of gemcitabine/cisplatin and panitumumab in patients with wild-type HRAS (non-mutated status). The progression-free survival rate at 12 months will be compared to expectations derived from historical data, which are verified by a randomised control group without the antibody.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, unresectable urothelial carcinoma of the bladder or the upper urinary tract
* Wild-type HRAS
* Male and female subjects > 18 years of age
* General condition ECOG 0-1
* Life expectancy at least 12 weeks
* Women of child-bearing potential: negative pregnancy test and use of effective contraception(oral contraceptive, coil); men: use of adequate male contraception (condom) for up to 3 months after discontinuation of panitumumab therapy
* Locally advanced or metastatic disease (T3b,T4 and/or N+ and/or M+)
* At least one unidimensionally measurable lesion detectable in CT or MRI corresponding to the RECIST criteria
* Adequate haematological, hepatic, renal and metabolic function parameters:

Leukocytes > 3000/mm³, ANC ≥ 1500/mm³, platelets ≥ 100,000/mm³, hemoglobin > 9 g/dl Creatinine clearance ≥ 50 ml/min and serum creatinine ≤ 1.5 x upper limit of normal Bilirubin ≤ 1.5 x upper limit of normal, GOT-GPT ≤ 2.5 x upper limit of normal in absence of liver metastases, or ≤ 5 x upper limit of normal in presence of liver metastases, AP ≤ 5 x upper limit of normal Magnesium ≥ lower limit of normal; calcium ≥ lower limit of normal INR and PTT < 1.5 x the upper limit of the normal reference range

Exclusion Criteria:

* HRAS mutation
* Absence of any of the above-listed inclusion criteria
* Dialysis-dependence following nephrectomy
* Patients with cerebral tumours and/or cerebral metastases
* Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrolment.
* Patients with uncontrolled hypertension; systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg despite optimal medical treatment
* History of interstitial lung disease, e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* Patients with thrombotic or embolic events, such as stroke or pulmonary embolism
* Patients with recent or known history of haemorrhagic diathesis
* Known significant neurological or psychiatric disorders, including dementia and epileptic seizures
* Serious inflammatory eye conditions, hearing impairment
* Pulmonary (pO2 < 60 mmHg), haemopoietic (e.g. serious bone marrow aplasia), hepatic or renal disorders
* Patients with poorly controlled diabetes mellitus
* Serious bacterial or fungal infections (>grade 2 NCI CTC Version 3)
* Chronic hepatitis B or C; HIV infection
* Autoimmune disease
* Allergic reaction to one of the medications to be used
* Status post organ transplantation
* Status post autologous bone marrow transplantation or stem cell transplantation in the 4 months prior to study commencement
* Manifest secondary malignancy or other form of cancer in the previous 5 years (excluding basalioma, in situ cervical cancer, incidental prostatic cancer)
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 3 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly).
* Active participation in other clinical studies in the previous 4 weeks
* Prior systemic therapy with cytostatics or immunotherapeutic agents
* Concurrent use of other anticancer treatments after study commencement
* Intravesical chemotherapy in the previous 4 weeks
* Radiotherapy in the previous 4 weeks
* Previous radiotherapy in which all lesions to be used for the evaluation of tumour response were irradiated
* Patients in a closed institution according to an authority or court decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Primary end point: Progression-free survival rate after 12 months. | 12 months

SECONDARY OUTCOMES:
Determination of best response (CR, PR and SD) rates in accordance with the RECIST criteria | up to 18 weeks
Duration of response, progression-free and overall survival time | 2 years
Documentation of adverse effects in accordance with the NCI CTC criteria | up to 18 weeks
Documentation of quality of life on the basis of the EORTC questionnaire | up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Miller, Prof. Dr., Principal Investigator — Universitätsmedizin Charité Berlin, Klinik für Urologie
Locations (20):
- Germany (20):
  - Bundeswehrkrankenhaus Berlin, Berlin
  - Krankenhaus am Urban, Berlin
  - Heilig-Geist-Krankenhaus, Cologne
  - St.-Josefs-Hospitals Dortmund, Dortmund
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum Fulda, Fulda
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Urologie, Hanover
  - Universitätskllinikum Heidelberg, Heidelberg
  - Klinikum Kassel, Kassel
  - Klinikum Ludwigshafen, Ludwigshafen
  - Universitätsklinikum Mainz, Mainz
  - Uroloische Praxis, Markkleeberg
  - Universitätsklinikum Münster, Münster
  - Johanniter Krankenhaus, Stendal
  - Universitätsklinikum Ulm, Urologische Klinik, Ulm
  - Klinikum Weiden, Weiden
  - Gemeinschaftspraxis für Urologie DGU, Wuppertal